CLINICAL TRIAL: NCT03791281
Title: Beliefs and Attitudes for Successful Implementation in Schools (BASIS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Aaron Lyon, Associate Professor, School of Medicine: Psychiatry: Childrens Division, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 52139; 1R21MH108714 (NIH)
Record Dates: First submitted 2018-12-21; First posted 2019-01-02 (Actual); Last update posted 2019-01-02 (Actual); Status verified 2018-12

CONDITIONS: Intervention Adoption; Implementation
Keywords: pre-implementation intervention; implementation strategy; individual-level barriers

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BASIS (Experimental): Received a 3-hour BASIS implementation strategy.
  Interventions: Behavioral: BASIS
- Attention Control (Active Comparator): Received a 3-hour session designed to control for dose, information provided, and presenter effects.
  Interventions: Behavioral: Attention Control

INTERVENTIONS:
Behavioral: BASIS
  Arms: BASIS
Behavioral: Attention Control
  Arms: Attention Control

SUMMARY:
The goal of this study is to adapt and test the feasibility and potential efficacy of a theory-driven pre-implementation intervention to address individual-level barriers to EBP implementation - Beliefs and Attitudes for Successful Implementation in Schools (BASIS) - designed to improve school mental health providers' implementation of EBPs. BASIS is intended to be a feasible and scalable first-line or adjunctive implementation enhancement intervention that is facilitative of other efforts (e.g., organizational interventions) that target high quality EBP implementation. Aims of this study are to: (1) Adapt an existing, theory-driven implementation intervention (BASIS), previously used with educators, to improve the EBP implementation behaviors of school mental health providers; and (2) Assess the viability of a later clinical trial by: (a) establishing the feasibility, acceptability, and appropriateness of the BASIS intervention among school mental health providers, and (b) Pilot testing BASIS, as compared to an Attention Control, delivered as pre-implementation intervention prior to training in a specific, existing EBP. Key organizational factors (e.g., implementation climate) will also be evaluated and included as covariates and we will explore trends in the data to inform the design of a larger trial. Ultimately, BASIS offers an innovative and scalable approach to improving school mental health providers' uptake and use of EBPs in order to increase the number of youth with mental health problems who receive high quality services.

ELIGIBILITY:
Inclusion:

School mental health providers (school psychologists, school social workers, etc.) recruited from middle and high schools in two economically and ethnically diverse districts in the Seattle area.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2016-08-15 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Change in Attitudes toward Evidence-Based Practices | Pre-intervention/baseline, post-intervention (1-2 weeks), 4-month follow-up
  Evidence-Based Practice Attitudes Scale (EBPAS) is a widely used 26-item tool designed to assess evidence-based practice (EBP) attitudes with items measured on a 0-4 scale and 6 subscales: (1) likelihood of adopting if the EBP were a requirement; (2) likelihood of adopting if the EBP were appealing to you; (3) openness to new practices; (4) perceived divergence between current practices and EBPs; (5) fit of EBPs with current practices; and (6) burden of EBPs. Subscale and total scores are mean scores of items with a range of 0-4. Higher scores reflect more favorable attitudes (perceived divergence is reverse-coded).
Change in Subjective Norms | Pre-intervention/baseline, post-intervention (1-2 weeks), 4-month follow-up
  Subjective Norms Scale is based on Theory of Planned Behavior (TPB) constructs. Two subscales measure two types implementation-related subjective norms: injunctive norms and descriptive norms. Four items load on each subscale and mean score range from -3 to +3, with positive scores reflecting more positive subjective injunctive and descriptive norms.
Change in Perceived Behavioral Control | Pre-intervention/baseline, post-intervention (1-2 weeks), 4-month follow-up
  Perceived Behavioral Control Scale is a modified version of the Teacher's Self-Efficacy Scale, which has 10 items assessing perceived behavioral control in implementing evidence-based practices. Items are scored on a 1-4 scale with a total mean score ranging from 1-4. Higher scores reflect greater (i.e., more favorable) perceived behavioral control.

SECONDARY OUTCOMES:
Change in School Implementation Citizenship Behaviors | Pre-intervention/baseline, post-intervention (1-2 weeks), 4-month follow-up
  The School Implementation Citizenship Behaviors Scale (S-ICBS) includes 15 items and measures clinicians' perceptions of how school staff engage with evidence-based practices in their specific school context. There are 4 subscales: (1) helping others; (2) keeping informed; (3) taking initiative; and (4) advocacy. Subscale and total scores are mean scores of items with a range of 0-4. Higher scores reflect greater (i.e., more favorable) implementation citizenship behavior.
Change in Intentions to Implement | Pre-intervention/baseline, post-intervention (1-2 weeks), 4-month follow-up
  The Modified Intentions to Use Scale has 9 items assessing school mental health providers' intentions to implement evidence-based practices. A total mean score is computed with a range of 0-4 and higher scores indicate more favorable intentions. Two versions of this scale were administered. At baseline, all providers were asked about general intentions to implement evidence-based practices. After training, clinicians were asked about intentions to implement the specific intervention for which they had received training.

CONTACTS AND LOCATIONS:
Overall Officials: Aaron R Lyon, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington School Mental Health Assessment, Research, and Training (SMART) Center, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lyon AR, Cook CR, Duong MT, Nicodimos S, Pullmann MD, Brewer SK, Gaias LM, Cox S. The influence of a blended, theoretically-informed pre-implementation strategy on school-based clinician implementation of an evidence-based trauma intervention. Implement Sci. 2019 May 30;14(1):54. doi: 10.1186/s13012-019-0905-3. PMID 31146788